CLINICAL TRIAL: NCT07120360
Title: Effect of Gender-Based Microaggression Awareness and Prevention Psychoeducation Program on Gender Role Attitudes and Gender Role Stress of Female University Students
Brief Title: Gender Microagression Psychoeducation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Kadriye Aslan, Graduate Student, Yuzuncu Yil University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/06-13
Record Dates: First submitted 2025-04-26; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Mental Health
Keywords: microaggression; mental health; Psychoeducation
MeSH Terms: conditions — Psychological Well-Being; Microaggression

STUDY DESIGN:
Intervention Model Description: This study evaluated a psychoeducation program comprising six modules, aiming to increase microaggression awareness, develop coping skills, enhance critical thinking on gender roles, and reduce gender role stress among female university students. The program included theoretical knowledge, experiential learning, assertiveness training, and stress management techniques. The sample included 80 female students, with 31 assigned to the experimental group and 49 to the control group. The experimental group received the full program, while the control group did not receive any intervention during the study but was given a brief educational session afterward. Data were collected at two points-pre-test and post-test-using the Personal Information Form, Ambivalent Sexism Inventory, Female Microaggression Scale, Depression Anxiety Stress Scale (DASS-21), and a semi-structured interview developed by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation Group (Experimental): Participants in this arm received a six-session psychoeducation program designed to increase awareness of gender-based microaggressions, develop coping and assertiveness skills, foster critical thinking regarding gender roles, and reduce gender role stress. The program included theoretical education, experiential learning exercises, group discussions, assertiveness training, and stress management strategies. Sessions were conducted face-to-face in small groups over a three-week period, with each session lasting approximately 60-90 minutes.
  Interventions: Other: Gender-Based Microaggression Awareness and Prevention Psychoeducation Program
- Control Group (No Intervention): No Intervention

INTERVENTIONS:
Other: Gender-Based Microaggression Awareness and Prevention Psychoeducation Program — The psychoeducation program consisted of six modules aiming to increase awareness of microaggressions, develop coping and assertiveness skills, enhance critical thinking regarding gender roles, and reduce gender role stress. The program included theoretical knowledge, experiential learning, assertiveness training, and stress management strategies.
  Arms: Psychoeducation Group

SUMMARY:
Objective: This study evaluates the effectiveness of the Gender-Based Microaggression Awareness and Prevention Psychoeducation Program, which was designed to enhance awareness of gender-based microaggressions among female university students and to improve their coping skills. The program's impact on gender role attitudes and psychological distress was also examined.

Methods: The research employed a quasi-experimental design with pre-test and post-test measurements. Gender-based microaggressions are defined as subtle but harmful actions or expressions targeting individuals' identities, often perpetrated unconsciously. In particular, gender-based microaggressions perpetuate traditional gender roles, undermine women's autonomy, and negatively affect psychological well-being, constituting invisible barriers in social and professional life.

The psychoeducation program consisted of six modules aiming to increase awareness of microaggressions, develop coping and assertiveness skills, enhance critical thinking regarding gender roles, and reduce gender role stress. The program included theoretical knowledge, experiential learning, assertiveness training, and stress management strategies. A total of 80 students participated, with 31 assigned to the experimental group and 49 to the control group.

Instruments: Data were collected using the Personal Information Form, Ambivalent Sexism Inventory, Female Microaggressions Scale, Depression-Anxiety-Stress Scale (DASS-21), and semi-structured interviews prepared by the researcher.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman,
* Knowing Turkish,
* Not having any communication problems (language, hearing, etc.).
* Being 18 years of age or older,
* Being willing to participate in the research.

Exclusion Criteria:

* Having a mental or physical problem that prevents communication,
* Being male

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Being female
Enrollment: 80 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Gender microagressions level | From enrollment to the end of psychoeducation at 6 weeks
  The scale developed by Miyake (2018) aims to measure gender-based microaggressions experienced by women throughout their lives. The scale was developed through a two-phase study and consists of eight thematic factors: sexual objectification; second-class citizenship/assumptions of inferiority; traditional gender roles; denial of sexism; sexist language use; environmental microaggressions; implicit threat to physical safety; and explicit threat to physical safety. Each factor represents a specific form of microaggression, using thematic classifications instead of the typical categories of microassaults, microinsults, or microinvalidations. The scale includes 34 items rated on a 4-point Likert scale (1 = Never, 4 = Often).
Gender Role Attitudes | From enrollment to the end of treatment at 6 weeks
  The Ambivalent Sexism Inventory (ASI) was developed by Glick and Fiske (1996) to assess perceptions of sexism and adapted into Turkish by Sakallı-Uğurlu (2002). The scale consists of 22 items rated on a 6-point Likert scale (1 = strongly disagree, 6 = strongly agree) and includes two subscales: hostile sexism and benevolent sexism. Hostile sexism reflects negative attitudes and discriminatory behaviors toward women, emphasizing their inferiority and weakness. Benevolent sexism involves seemingly positive but patronizing attitudes based on patriarchal values, such as the belief that women should be protected and cherished. Although conceptually distinct, both dimensions contribute to the persistence of gender inequality. Higher scores indicate higher levels of hostile or benevolent sexism.
Psychological Distress Level | From enrollment to the end of treatment at 6 weeks
  The Depression Anxiety Stress Scales (DASS) were developed by Lovibond and Lovibond (1995) to assess three components of negative emotional states: depression, anxiety, and stress. The original scale includes 42 items rated on a 4-point Likert scale (0 = Did not apply to me at all, 3 = Applied to me very much). The short version, DASS-21, was developed by Antony et al. (1998) and has been shown to be a valid and reliable tool. The Turkish adaptation of DASS-21 was conducted by Sarıçam (2018). The scale does not produce a total score; instead, each subscale is scored separately, with scores ranging from 0 to 21. Higher scores indicate higher levels of depression, anxiety, or stress in the corresponding subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Cemile H AYHAN, Assoc. Prof., Study Director — Yuzuncu Yil University; Kadriye ASLAN, Graduate student, Principal Investigator — Yuzuncu Yil University
Locations (2):
- Turkey (Türkiye) (2):
  - Van Yuzuncu Yıl University Campus /Faculty of Health Sciences/van/turkey, Van, Tusba
  - Van Yuzuncu Yıl University, Van, Tusba

IPD SHARING:
Plan to Share IPD: No
I won't share thanks

REFERENCES:
- [Background] Turner J, Higgins R, Childs E. Microaggression and Implicit Bias. Am Surg. 2021 Nov;87(11):1727-1731. doi: 10.1177/00031348211023418. Epub 2021 Jun 2. PMID 34078131
- [Background] Sue DW, Capodilupo CM, Torino GC, Bucceri JM, Holder AM, Nadal KL, Esquilin M. Racial microaggressions in everyday life: implications for clinical practice. Am Psychol. 2007 May-Jun;62(4):271-86. doi: 10.1037/0003-066X.62.4.271. PMID 17516773
- [Background] Marchi M, Travascio A, Uberti D, De Micheli E, Quartaroli F, Laquatra G, Grenzi P, Pingani L, Ferrari S, Fiorillo A, Converti M, Pinna F, Amaddeo F, Ventriglio A, Mirandola M, Galeazzi GM. Microaggression toward LGBTIQ people and implications for mental health: A systematic review. Int J Soc Psychiatry. 2024 Feb;70(1):23-35. doi: 10.1177/00207640231194478. Epub 2023 Aug 28. PMID 37638668
- See also: Related Info — https://scholar.google.com/scholar?hl=tr&as_sdt=0%2C5&q=gender+microaggressions&oq=gender+micr